CLINICAL TRIAL: NCT00227435
Title: A Phase I/II Double-Blind, Dose Escalation Study to Evaluate the Safety, Pharmacokinetics and Antiviral Activity of Val-mCyd (NM283) in Adults With Chronic Hepatitis C
Brief Title: Dose Escalation Study to Evaluate the Safety and Antiviral Activity of Val-mCyd in Adults With Chronic Hepatitis C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV-08A-001
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

INTERVENTIONS:
Drug: val-mCyd

SUMMARY:
This study was conducted to determine the safety, tolerance, pharmacokinetics and antiviral activity of val-mCyd at doses ranging from 50 mg to 800 mg per day.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical history of chronic hepatitis C and compensated liver disease
* No antiviral treatment for hepatitis C in the 6 months prior to the Screening visit

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co-infected with HBV or HIV

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Pasadena, California
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Fairfax, Virginia